CLINICAL TRIAL: NCT04127071
Title: Study Protocol for A Randomized Controlled Trial of Incision and Drainage Versus Ultrasound-Guided Needle Aspiration for Uncomplicated Skin Abscesses
Brief Title: Abscess Aspiration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Robert Ehrman, Assistant Professor of Emergency Medicine, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1804001385
Record Dates: First submitted 2019-10-10; First posted 2019-10-15 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Skin Abscess
Keywords: Ultrasound Guided Needle Aspiration; Incision and Drainage
MeSH Terms: conditions — Surgical Wound | interventions — Drainage

STUDY DESIGN:
Intervention Model Description: A prospective, nonblinded, randomized controlled trial comparing ultrasound-guided needle aspiration to incision and drainage of uncomplicated skin abscesses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical I&D Procedure (Active Comparator): The abscess cavity will be evaluated thoroughly with ultrasonography. The site will be prepared and draped. The skin surface will be infiltrated with local anesthetic with a 25-gauge needle. The treating clinician may provide ultrasound-guided regional anesthesia for procedural analgesia at their discretion. Incision of the skin surface with a number 11-blade scalpel will be performed over the largest area of infection; the incision will be extended into the abscess cavity. A blunt instrument will then be used to break up internal loculations if present. Repeated instrumentation through the initial incision or extension of the original incision will be performed if needed. Lastly, iodoform packing will be inserted through the incision into the cavity. The decision to send the abscess contents for microbiological culture and susceptibility analysis will be at the discretion of the treating clinician.
  Interventions: Procedure: Incision and Drainage (I&D)
- Ultrasound-guided Needle Aspiration Procedure (Experimental): The abscess cavity will be evaluated thoroughly with US. The site will be prepared and draped. The skin surface and anticipated needle track will be infiltrated with local anesthetic with a 25g needle. The treating clinician may provide ultrasound-guided regional anesthesia for procedural analgesia at their discretion. Under direct US-guided visualization, a 14g 2in steel needle attached to a 40mL syringe will be advanced into the abscess cavity with manual negative pressure. The needle tract will be extended obliquely 2-3 cm between the skin and abscess to prevent fistulization. Purulent material will be aspirated until no further purulence can be aspirated. Multiple aspiration attempts on the initial visit will be permitted to maximally drain the abscess cavity. Additionally, irrigation of the abscess cavity with sterile saline will be permitted to break up internal loculations if present, as has reported previously for trunk and breast abscesses.
  Interventions: Procedure: Ultrasound-guided Needle Aspiration Procedure

INTERVENTIONS:
Procedure: Ultrasound-guided Needle Aspiration Procedure — The intervention under investigation utilizes an ultrasound-guided needle to less invasively drain an abscess.
  Arms: Ultrasound-guided Needle Aspiration Procedure
Procedure: Incision and Drainage (I&D) — The current standard procedure to drain an abscess of purulent material.
  Arms: Surgical I&D Procedure

SUMMARY:
Incision and drainage (I&D) is the standard guideline treatment of uncomplicated skin abscesses (a boil or bumo beneath the skin). Ultrasound-guided needle aspiration (USGNA) is a minimally invasive and less painful alternative treatment, but has not been validated as non-inferior to I&D. Multiple studies have shown successful treatment with USGNA of breast, face, neck, and/or trunk abscesses in combination with oral antibiotics with success rates as high as 97%.

In 2011 Gaspari et al. published a landmark article on the use of USGNA for skin abscesses. In this randomized controlled trial, USGNA and I&D had failure rates of 74% and 20% respectively, which makes USGNA an unappealing treatment option. However, the study had several methodological issues that likely biased the results in favor of I&D, including the following: 1) aspiration was performed with an 18-gauge needle which is often too small to aspirate thick purulence (or pus); 2) failure to fully aspirate all abscess contents was a priori defined as treatment failure rather than strictly clinical outcomes; 3) the abscess aspiration procedure was not standardized; and 4) post-intervention oral antibiotic therapy was not used on all patients.

The main hypothesis is that a modified protocol of the Gaspari et al. USGNA study to address these flaws will demonstrate a failure of USGNA comparable to I&D for the treatment of uncomplicated skin abscesses. First, the study will standardize the use of larger 14-gauge needle on all USGNAs. Second, USGNA intervention failure need not be defined as the inability to completely aspirate all abscess cavity contents under ultrasound guidance. Previous studies have demonstrated clinical success with USGNA of skin abscesses without applying the rigid failure criteria chosen by Gaspari et al. There is only one study in the literature to suggest that there is no correlation between a small quantity of residual abscess contents post-USGNA and ultimate clinical failure, however, there are no studies which specifically address this clinical question. In this study, initial treatment failure of USGNA will be defined as the inability to aspirate any purulent material. Third, treatment outcomes in this study will be determined by clinical resolution of abscess at the study endpoint of 7-10 days, which is a well-established timeline for anticipated abscess healing and endpoint clinical follow-up. Fourth, ultrasound fellowship-trained emergency physicians will perform USGNA in standardized fashion on all enrolled patients. Lastly, post-intervention oral antibiotic with methicillin-resistant Staphylococcus aureus (MRSA) coverage will be provided and compliance closely monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Non-toxic patients who present with an uncomplicated, superficial skin abscess of the head/neck, torso, extremities, and buttock will be eligible for inclusion.
2. Abscesses must be verified by physical examination and bedside ultrasound.
3. Patients with clinical history of diabetes mellitus and previous diagnosis of MRSA will be included.

Exclusion Criteria:

1. Patients will be excluded if age less than age 18 or pregnant.
2. Patient or legal guardian is unable to give consent.
3. Patients with no means of clinical follow-up will be excluded.
4. Complicated abscesses, defined as an abscess with associated sepsis, lymphangitis, or osteomyelitis, requiring intravenous antibiotic therapy, requiring hospital admission, previous surgical drainage at site of abscess, overlying skin lesion/fistula/ulceration with the exception of cellulitis, perforated or actively draining abscess, duration of symptoms > 5 days,1,28 and/or multiple concurrent abscesses that can be clinically regarded as chronic in nature will be excluded.

4) Abscess locations which will be excluded are dental, peritonsillar, anorectal, genital/inguinal, axillary if suspicion for chronic hidradenitis suppurativa, or pilonidal/intragluteal at the base of the coccyx.

5) Abscesses greater in size than 3x3x3 cm in any dimension will be excluded. [It has been suggested extensively in the surgical literature that an abscess diameter >3 cm should have surgical/catheter-drainage as the initial management instead of needle aspiration]2,5,15,19,27,33 [It has been reported that abscesses >3 cm in size have increased failure rates]15 6) Abscess depth is greater than maximal needle length. 7) Patients with immunosuppression from following clinical conditions will be excluded: HIV, cancer on active chemotherapy.

8) Patients with active history of IV drug use will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Abscess cure or treatment failure | 7-10 days
  Treatment cure will be defined by the complete resolution of the abscess based on clinical signs and symptoms (no or minimal tenderness, erythema, fever, wound drainage, warmth, fluctuance, or induration) at the 7- to 10-day follow-up. Treatment failure will be defined by: fever (attributable to the infection), persistent or increased size >25% of the original abscess, requiring conversion to I&D (USGNA intervention group) or repeat I&D (I&D intervention group), requiring additional antibiotics, or requiring hospital admission within 7-10 days after treatment. Participants who either withdraw from the trial or are lost to follow-up before a determination of final outcome will be classified as treatment failure.

SECONDARY OUTCOMES:
Patient Satisfaction | Baseline (Day 1)
  Patient satisfaction with each procedural intervention will be assessed, with the hypothesis that USGNA will have higher overall satisfaction rates than I&D.
Patient Comfort Level | Baseline (Day 1)
  Patient comfort for each procedural intervention will be assessed , with the hypothesis that USGNA will have lower overall pain scores compared to I&D.
Abscess Characteristics and Correlation with Treatment Failure | Baseline (Day 1)
  Assessment of whether specific abscess characteristics have any correlation to procedural failure in either intervention group.
Abscess Reoccurrence | Day 21-30
  The cumulative rate of abscess recurrence will be assessed at the 21- to 30-day follow-up.
Abscess Site infection | Day 21-30
  Infections involving the same site at the 21- to 30-day follow-up will be considered a recurrent infection.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ehrman, MD, Principal Investigator — Wayne State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barron AU, Luk S, Phelan HA, Williams BH. Do acute-care surgeons follow best practices for breast abscess management? A single-institution analysis of 325 consecutive cases. J Surg Res. 2017 Aug;216:169-171. doi: 10.1016/j.jss.2017.05.013. Epub 2017 May 10. PMID 28807202
- [Background] Berna-Serna JD, Madrigal M, Berna-Serna JD. Percutaneous management of breast abscesses. An experience of 39 cases. Ultrasound Med Biol. 2004 Jan;30(1):1-6. doi: 10.1016/j.ultrasmedbio.2003.10.003. PMID 14962601
- [Background] Blaivas M. Ultrasound-guided breast abscess aspiration in a difficult case. Acad Emerg Med. 2001 Apr;8(4):398-401. doi: 10.1111/j.1553-2712.2001.tb02122.x. PMID 11282679
- [Background] Chandika AB, Gakwaya AM, Kiguli-Malwadde E, Chalya PL. Ultrasound Guided Needle Aspiration versus Surgical Drainage in the management of breast abscesses: a Ugandan experience. BMC Res Notes. 2012 Jan 6;5:12. doi: 10.1186/1756-0500-5-12. PMID 22226127
- [Background] Christensen AF, Al-Suliman N, Nielsen KR, Vejborg I, Severinsen N, Christensen H, Nielsen MB. Ultrasound-guided drainage of breast abscesses: results in 151 patients. Br J Radiol. 2005 Mar;78(927):186-8. doi: 10.1259/bjr/26372381. PMID 15730981
- [Background] Chuck EA, Frazee BW, Lambert L, McCabe R. The benefit of empiric treatment for methicillin-resistant Staphylococcus aureus. J Emerg Med. 2010 Jun;38(5):567-71. doi: 10.1016/j.jemermed.2007.11.037. Epub 2008 Jun 2. PMID 18514468
- [Background] Dixon JM. Repeated aspiration of breast abscesses in lactating women. BMJ. 1988 Dec 10;297(6662):1517-8. doi: 10.1136/bmj.297.6662.1517. No abstract available. PMID 3147056
- [Background] Dixon JM. Outpatient treatment of non-lactational breast abscesses. Br J Surg. 1992 Jan;79(1):56-7. doi: 10.1002/bjs.1800790120. PMID 1737278
- [Background] Elagili F, Abdullah N, Fong L, Pei T. Aspiration of breast abscess under ultrasound guidance: outcome obtained and factors affecting success. Asian J Surg. 2007 Jan;30(1):40-4. doi: 10.1016/S1015-9584(09)60126-3. PMID 17337370
- [Background] Frazee BW, Lynn J, Charlebois ED, Lambert L, Lowery D, Perdreau-Remington F. High prevalence of methicillin-resistant Staphylococcus aureus in emergency department skin and soft tissue infections. Ann Emerg Med. 2005 Mar;45(3):311-20. doi: 10.1016/j.annemergmed.2004.10.011. PMID 15726056
- [Background] Garg P, Rathee SK, Lal A. Ultrasonically guided percutaneous drainage of breast abscess. J Indian Med Assoc. 1997 Nov;95(11):584-5. PMID 9567588
- [Background] Gaspari RJ, Resop D, Mendoza M, Kang T, Blehar D. A randomized controlled trial of incision and drainage versus ultrasonographically guided needle aspiration for skin abscesses and the effect of methicillin-resistant Staphylococcus aureus. Ann Emerg Med. 2011 May;57(5):483-91.e1. doi: 10.1016/j.annemergmed.2010.11.021. Epub 2011 Jan 15. PMID 21239082
- [Background] Giess CS, Golshan M, Flaherty K, Birdwell RL. Clinical experience with aspiration of breast abscesses based on size and etiology at an academic medical center. J Clin Ultrasound. 2014 Nov-Dec;42(9):513-21. doi: 10.1002/jcu.22191. Epub 2014 Jun 27. PMID 24975466
- [Background] Herzon FS. Needle aspiration of nonperitonsillar head and neck abscesses. A six-year experience. Arch Otolaryngol Head Neck Surg. 1988 Nov;114(11):1312-4. doi: 10.1001/archotol.1988.01860230106035. PMID 3166766
- [Background] Hook GW, Ikeda DM. Treatment of breast abscesses with US-guided percutaneous needle drainage without indwelling catheter placement. Radiology. 1999 Nov;213(2):579-82. doi: 10.1148/radiology.213.2.r99nv25579. PMID 10551245
- [Background] Imperiale A, Zandrino F, Calabrese M, Parodi G, Massa T. Abscesses of the breast. US-guided serial percutaneous aspiration and local antibiotic therapy after unsuccessful systemic antibiotic therapy. Acta Radiol. 2001 Mar;42(2):161-5. doi: 10.1080/028418501127346666. PMID 11259943
- [Background] Kang YD, Kim YM. Comparison of needle aspiration and vacuum-assisted biopsy in the ultrasound-guided drainage of lactational breast abscesses. Ultrasonography. 2016 Apr;35(2):148-52. doi: 10.14366/usg.15041. Epub 2015 Dec 8. PMID 26753603
- [Background] Karstrup S, Nolsoe C, Brabrand K, Nielsen KR. Ultrasonically guided percutaneous drainage of breast abscesses. Acta Radiol. 1990 Mar;31(2):157-9. PMID 2196923
- [Background] Karstrup S, Solvig J, Nolsoe CP, Nilsson P, Khattar S, Loren I, Nilsson A, Court-Payen M. Acute puerperal breast abscesses: US-guided drainage. Radiology. 1993 Sep;188(3):807-9. doi: 10.1148/radiology.188.3.8351352.
- [Background] Kjaer S, Rud B, Bay-Nielsen M. Ultrasound-guided drainage of subcutaneous abscesses on the trunk is feasible. Dan Med J. 2013 Apr;60(4):A4601. PMID 23651712
- [Background] Leborgne F, Leborgne F. Treatment of breast abscesses with sonographically guided aspiration, irrigation, and instillation of antibiotics. AJR Am J Roentgenol. 2003 Oct;181(4):1089-91. doi: 10.2214/ajr.181.4.1811089. PMID 14500237
- [Background] May L, Harter K, Yadav K, Strauss R, Abualenain J, Keim A, Schmitz G. Practice patterns and management strategies for purulent skin and soft-tissue infections in an urban academic ED. Am J Emerg Med. 2012 Feb;30(2):302-10. doi: 10.1016/j.ajem.2010.11.033. Epub 2011 Jan 28. PMID 21277138
- [Background] May LS, Zocchi M, Zatorski C, Jordan JA, Rothman RE, Ware CE, Eells S, Miller L. Treatment Failure Outcomes for Emergency Department Patients with Skin and Soft Tissue Infections. West J Emerg Med. 2015 Sep;16(5):642-52. doi: 10.5811/westjem.2015.7.26213. Epub 2015 Oct 20. PMID 26587085
- [Background] Moran GJ, Krishnadasan A, Gorwitz RJ, Fosheim GE, McDougal LK, Carey RB, Talan DA; EMERGEncy ID Net Study Group. Methicillin-resistant S. aureus infections among patients in the emergency department. N Engl J Med. 2006 Aug 17;355(7):666-74. doi: 10.1056/NEJMoa055356. PMID 16914702
- [Background] O'Hara RJ, Dexter SP, Fox JN. Conservative management of infective mastitis and breast abscesses after ultrasonographic assessment. Br J Surg. 1996 Oct;83(10):1413-4. doi: 10.1002/bjs.1800831028. PMID 8944458
- [Background] Olderog CK, Schmitz GR, Bruner DR, Pittoti R, Williams J, Ouyang K. Clinical and epidemiologic characteristics as predictors of treatment failures in uncomplicated skin abscesses within seven days after incision and drainage. J Emerg Med. 2012 Oct;43(4):605-11. doi: 10.1016/j.jemermed.2011.09.037. Epub 2012 Jun 12. PMID 22698825
- [Background] Ozseker B, Ozcan UA, Rasa K, Cizmeli OM. Treatment of breast abscesses with ultrasound-guided aspiration and irrigation in the emergency setting. Emerg Radiol. 2008 Mar;15(2):105-8. doi: 10.1007/s10140-007-0683-0. Epub 2008 Jan 10. PMID 18193464
- [Background] Schwarz RJ, Shrestha R. Needle aspiration of breast abscesses. Am J Surg. 2001 Aug;182(2):117-9. doi: 10.1016/s0002-9610(01)00683-3. PMID 11574080
- [Background] Singer AJ, Talan DA. Management of skin abscesses in the era of methicillin-resistant Staphylococcus aureus. N Engl J Med. 2014 Mar 13;370(11):1039-47. doi: 10.1056/NEJMra1212788. No abstract available. PMID 24620867
- [Background] Stevens DL, Bisno AL, Chambers HF, Dellinger EP, Goldstein EJ, Gorbach SL, Hirschmann JV, Kaplan SL, Montoya JG, Wade JC. Practice guidelines for the diagnosis and management of skin and soft tissue infections: 2014 update by the infectious diseases society of America. Clin Infect Dis. 2014 Jul 15;59(2):147-59. doi: 10.1093/cid/ciu296. Epub 2014 Jun 18. PMID 24947530
- [Background] Talan DA, Mower WR, Krishnadasan A, Abrahamian FM, Lovecchio F, Karras DJ, Steele MT, Rothman RE, Hoagland R, Moran GJ. Trimethoprim-Sulfamethoxazole versus Placebo for Uncomplicated Skin Abscess. N Engl J Med. 2016 Mar 3;374(9):823-32. doi: 10.1056/NEJMoa1507476. PMID 26962903
- [Background] Tan SM, Low SC. Non-operative treatment of breast abscesses. Aust N Z J Surg. 1998 Jun;68(6):423-4. doi: 10.1111/j.1445-2197.1998.tb04791.x. PMID 9623462
- [Background] Ulitzsch D, Nyman MK, Carlson RA. Breast abscess in lactating women: US-guided treatment. Radiology. 2004 Sep;232(3):904-9. doi: 10.1148/radiol.2323030582. Epub 2004 Jul 29. PMID 15284435
- [Background] Yusa H, Yoshida H, Ueno E, Onizawa K, Yanagawa T. Ultrasound-guided surgical drainage of face and neck abscesses. Int J Oral Maxillofac Surg. 2002 Jun;31(3):327-9. doi: 10.1054/ijom.2002.0233. PMID 12190142